CLINICAL TRIAL: NCT05486624
Title: The Effect of Reiki Application Episiotomy Recovery and Perineal Pain
Brief Title: The Effect of Reiki Application on Episiotomy and Perineal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Halime AYDEMİR, Faculty of Health Sciences / Midwifery Department / Assistant Professor Doctor, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AhiEvranU
Record Dates: First submitted 2022-06-30; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Episiotomy; Birth; Perineal Pain
Keywords: Reiki; episiotomy; perineal pain; puerparant
MeSH Terms: interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: 1 control group, 1 intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Introductory Information Form was used in the control group on the 1st day of birth with face-to-face interviews. REEDA Scale, MAI-SF were used on the 1st, 2nd, 7th and 14th days of delivery. On the 1st day of birth, the Episiotomy Care Education Brochure and the Follow-up Form to be filled in within 14 days and to be obtained from them at the last follow-up were given. control group; It was evaluated by making a home visit on the 1st day and the 2nd day in the hospital, and on the 7th and 14th days. The records of the forms were filled by the researcher. Data collection time took approximately 15 minutes for the control group. Reiki was not applied to this group.
- Intervention group (Experimental): Introductory Information Form was used in the intervention group on the 1st day of birth with face-to-face interviews. REEDA Scale, MAI-SF were used on the 1st, 2nd, 7th and 14th days of delivery. On the 1st day of birth, the Episiotomy Care Education Brochure and the Follow-up Form to be filled in within 14 days and to be obtained from them at the last follow-up were given. intervention group; It was evaluated by making a home visit on the 1st day and the 2nd day in the hospital, and on the 7th and 14th days. Reiki was applied on the 1st, 2nd and 7th days of birth. In total, 3 sessions of Reiki were applied. The records of the forms were filled by the researcher. Data collection took approximately 50-55 minutes for the intervention group.
  Interventions: Other: Reiki

INTERVENTIONS:
Other: Reiki — Reiki, one of the complementary treatments, was applied by touching the chakra areas of the body by hand.
  Arms: Intervention group

SUMMARY:
Purpose: To investigate the effect of Reiki application on postpartum episiotomy recovery and perineal pain in postpartum women who had vaginal delivery.

Design and framework: The research is randomized controlled in a pre-test post-test order in a hospital in Turkey. By using Simple Random Numbers Table as the randomization method in the selection of the sample, a total of 86 puerperal women, 40 in the intervention group and 46 in the control group, were recruited. Episiotomy recovery of the intervention and control groups on the 1st day, 2nd day, 7th day, and 14th day postpartum was evaluated with the REEDA Scale, and perineal pain was evaluated with the McGill Pain Scale Short Form.

Participants: Postpartum women who gave vaginal birth participated in the study.

Intervention: 3 sessions of Reiki for 35-40 minutes were applied to the intervention group on the 1st, 2nd and 7th days of birth.

Results: There was a significant difference between the mean REEDA Scale edema scores in the 7th day (p=0.028) and 14th day (p=0.013) follow-up of the intervention and control groups. A significant difference was found between the 3rd post-test McGill Pain Scale Short Form total pain score averages (p=0.005) and the 4th follow-up McGill Pain Scale Short Form total pain score averages (p=0.001) of the intervention and control groups.

DETAILED DESCRIPTION:
The research is randomized controlled in the pre-test post-test order. This research has been reported in accordance with the CONSORT (Consolidated Standards of Reporting Trials) guidelines. Before working at the hospital, ethics committee approval (Number: 99166796-050.06.04) from Ege University Faculty of Medicine Dean's Medical Research Ethics Committee and institutional permission from Kırşehir Governorship Provincial Health Directorate Kırşehir Public Hospitals Services Unit (No: 42884709-806.99). The aim and content of the research were explained to the puerperants orally. In addition, verbal and written consent was obtained from the puerperants using the Informed Voluntary Consent Form. Postpartum women were informed that they have the right to leave the study whenever they want.

Randomization Simple Random Numbers Table was used as the randomization method in the sample selection of the study. Among the puerperant women who met the initial inclusion criteria, those who accepted to participate in the study were included in the application of randomization. Then, a randomly sorted algorithm was created at the maximum allowed percentage, with a deviation of 10%, in a total of 100 samples. In the algorithm, 50 sample (postpartum) groups for both groups; Up to 100 randomly sorted as A and B. Intervention group: A, Control group: B. The sample taken according to the order in the list on the data collection days; It is accepted as group A or B. In terms of equality according to the number of births of the groups, 50 sample groups were randomly divided into 2 groups of 25 each without being randomized. Two groups were formed as 25 puerperant primiparous group and 25 puerperal multiparous group. In the study, since the numbers in the multiparous group were completed earlier than in the primiparous group, the sampling was continued until the number of the primiparous group was completed.

Participants and Framework The smallest sample size to be taken in the research; In order to find the significant difference between the groups, repeated measurement variance analysis was determined by using Power (Gpower) analysis under the test. In the analysis, α=0.05 and f=0.25 (medium effect size) were taken with 80% power, and 78 cases were found to be sufficient. Considering the loss of follow-up, the number of samples was increased to 100. A total of 100 puerperant women, 50 puerperant women for each group, were included in the study. When the sample size was 100 cases, the power of analysis was checked again. The strength of the work "G. Calculated using the "Power-3.1.9.2" program. As a result of the analysis applied to 86 people, 40 in the intervention group and 46 in the control group, α = 0.05, the effect size was found to be 0.7882, and the power of the study, which was calculated as post-hoc, was calculated as 0.95. Patients aged 18 and over, no risky pregnancy (no systemic disease, no smoking, no postpartum complications), 37-42 weeks of gestation, single and live vaginal delivery, performed mediolateral episiotomy, no vaginal infection, any drug Postpartum women who do not use, do not have any laceration (anal sphincter injury, 3rd degree perineal laceration) other than episiotomy, use only clean water for perineal care and keep them dry are included. The puerperant women who had lacerations other than episiotomy, who did not meet the standards of using clean water in perineum care and keeping them dry (doing different care or using pharmacological products), and who did not accept home visits were excluded from the study. Out of 100 puerperant women included in the sample, although they initially accepted the home visit, 8 of them could not be reached for home visits, 3 of them were out of the province on the day of the home visit, 2 of them did not accept home visits, and 1 of them did not comply with the standard in perineal care. In the 4th follow-up, no home visit was made. In the intervention group; 10 puerperant women, 7 from the primiparous group and 3 from the multiparous group, did not complete the study. In the control group; 4 puerperant women, 2 from the primiparous group and 2 from the multiparous group, did not complete the study. Before the research, a pilot study was conducted with 12 puerperal women. The puerperant women taken in the pilot study were not included in the sample.

Introductory Information Form was used in the intervention and control groups on the 1st day of delivery by face-to-face interviews with the postpartum in the hospital. REEDA Scale, MAI-SF were used on the 1st, 2nd, 7th and 14th days of delivery in both groups. Both groups were given the Episiotomy Care Training Brochure on the 1st day of birth and the Follow-up Form, which they would fill in within 14 days and be taken from them at the last follow-up. Intervention and control group; It was evaluated by making a home visit on the 1st day and the 2nd day in the hospital, and on the 7th and 14th days. The records of the forms were filled by the researcher. Data collection time took approximately 15 minutes for the control group and approximately 50-55 minutes for the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* No risky pregnancy (no systemic disease, no smoking, no postpartum complications),
* The gestational week is 37-42 weeks,
* Single and live vaginal delivery,
* Mediolateral episiotomy performed,
* No vaginal infection,
* Not using any medication,
* No laceration (anal sphincter injury, 3rd degree perineal laceration) other than episiotomy,
* Only puerperant women who use clean water for perineum care and keep them dry will be included in the study.

Exclusion Criteria:

* Under 18 years old,
* Having a risky pregnancy,
* Gestational week other than 37-42 weeks,
* Having multiple births, stillbirths and anomalies,
* Having episiotomy other than mediolateral episiotomy,
* Having vaginal infection,
* Using any medication,
* Having laceration other than episiotomy,
* Cesarean section,
* Does not meet the standard of using clean water and keeping it dry in perineum care (doing different care or using pharmacological products),
* Postpartum women who do not accept home visits will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Sample power calculation | Before starting the research, power analysis was calculated.
  It is aimed to determine the number that will represent the universe by calculating the sample power in the study.
Introductory Information Form | 14 day
  In data collection, an Introductory Information Form consisting of 32 questions was used, which included information on socio-demographic characteristics, factors affecting wound healing, obstetric characteristics and hygiene characteristics of puerperant women.
REEDA Scale | 14 day
  The REEDA Scale was used by Davidson in 1974. The Turkish validity and reliability study was carried out using the specialty thesis on "The Effect of Hot and Cold Applications on Episiotomy Healing". The scale includes five factors that indicate perineal healing: redness, edema, ecchymosis, discharge, and approaching wound edges. Each improvement factor is evaluated by giving 0, 1, 2 and 3 points. The sum of the scores obtained as a result of the evaluation of five categories constitutes the REEDA score. The lowest score on the scale is 0, and the highest score is 15. The highest score on the scale indicates severe perineal trauma.
McGill Pain Scale Short Form (MAS-SF) | 14 day
  MAI-SF, developed by Melzack (1987), provides information about the sensory characteristics of pain, the severity of pain and the effect of pain. The Turkish validity and reliability of the MAI-SF has three parts. In the first part; There are 15 descriptive word groups and expressions containing the characteristics of pain. Descriptive words in this section are rated on an intensity scale from 0 to 3 (0 = none, 1 = mild, 2 = moderate, 3 = excessive). In the first part; A total of three pain scores are obtained: sensory pain score, perceptual pain score and total pain score. The sensory pain score is between 0-33 points, the perceptual pain score is between 0-12 points, and the total pain score is between 0-45 points. An increase in the score indicates an increase in pain. In the second part; There are five word groups ranging from "mild pain" to "unbearable pain" to determine the severity of pain. in the third part; Pain intensity is assessed using a 0-10 visual comparison scale.
Tracking Form | 14 day
  It is a form in which the 14-day follow-up of postpartum women is made. The status of using analgesics in the form, if he has taken analgesic drug, how many he has taken, how much time has passed between analgesic drugs, analgesic drug name-dose, breastfeeding status of the baby, breastfeeding frequency if he is breastfeeding, giving water/additional nutrition to his baby, and any other factors other than water in episiotomy care. There is information questioning the application status. It was given to the intervention and control groups at the first follow-up and was withdrawn at the fourth follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: NERİMAN S, Study Chair — neriman.sogukpinar@ege.edu.tr
Locations (1):
- Kırşehir Training and Research Hospital, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Billot, M, Daycard, M, Wood, C, Tchalla, A,. 2019. Reiki therapy for pain, anxiety and quality of life. BMJ Supportive & Palliative Care 9 (4), 434-438 — http://dx.doi.org/10.1136/bmjspcare-2019-001775
- See also: Chan, DW,. 2003. Hardiness and its role in the stres-burnout relationship among prospective Chinese teachers in Hong Kong. Teaching and Teacher Education 19 (4), 381-395 — https://doi.org/10.1016/S0742-051X(03)00023-4
- See also: World Health Organization. 2017. Recommendatıons On Maternal Health Guidelines Approved By The Who Guıdelines Review Committee Updated — http://apps.who.int/iris/bitstream/10665/259268/1/WHOMCA-17.10-eng.pdf
- See also: Royal College of Obstetricians and Gynaecologists (RCOG). 2021. Episiotomy — https://www.rcog.org.uk/en/patients/tears/episiotomy